CLINICAL TRIAL: NCT02370472
Title: Evaluation of a New Training Model for Ultrasound Guided Regional Anesthesia - A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Sanjib Adhikary, Associate Professor , Director Acute Pain, Regional Anesthesia/Orthopedics, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 38067
Record Dates: First submitted 2015-02-18; First posted 2015-02-25 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Regional Anesthesia
Keywords: Ultrasound; Image; Learning Tool; Ultrasound Guide Procedures; Simulated Setting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (No Intervention): complete pre-study form 10 minute familiarization time with equipment view video demonstration of task perform task 3 times assessed using scoring form - pretest assigned to group practice task again for 30 minutes proficiency noted final evaluation
- Experimental (Experimental): complete pre-study form 10 minute familiarization time with equipment view video demonstration of task perform task 3 times assessed using scoring form - pretest assigned to group practice task again for 30 minutes - subjects will use tool developed using cameras and a computer to visualize hand and needle movements as well as the position of the transducers along with the image from the ultrasound on a computer screen proficiency belief noted final evaluation
  Interventions: Other: tool developed using cameras and a computer

INTERVENTIONS:
Other: tool developed using cameras and a computer — cameras allowing subject to be able to visualize hand and needle movements as well s the position of the transducers along with the image from the ultrasound on a computer screen
  Arms: Experimental

SUMMARY:
The use of Ultrasound Guided Regional Anaesthesia (USRA) has increased over the last decade. Theoretically, ultrasound imaging may increase efficacy and safety by allowing visualization of the needle pathway and local anaesthetic spread around the nerve. In addition to knowledge of anatomy and general principles of ultrasonography, USRA requires learning new skills such as image interpretation, needle-beam alignment, and needle trajectory tracking. The hand-eye coordination required during needle advancement requires practice to master because the needle must be properly aligned with the ultrasound probe in order to maintain the needle path in the beam at all times. Adding to the difficulty, hand and needle movements can occur in three axes, but an ultrasound image is seen in only two dimensions. Since the ability to acquire the necessary skills to perform USRA is subjective and not yet validated, it is difficult to recommend a single, effective training pathway.

Currently, the only method of supervised training before performing an USRA procedure on an actual patient involves practicing needle insertion in a phantom or cadaver. Studies assessing the impact of learning using these methods are lacking. It is possible that some practitioners may choose alternative one-off learning methods. Such methods are not standardized and are thus difficult to evaluate.

DETAILED DESCRIPTION:
This was a single site, prospective, pre-test-post-test, randomized study conducted after Institutional Review Board (IRB) approval. Thirty subjects, including medical students, practicing anaesthesiologists and anaesthesia residents in training at the Penn State Hershey Medical Center, were recruited by formal email invitation to participate. Written consent was obtained from each participant before their inclusion in the study and each participant completed a pre-study form. Once enrolled in the study, participants were given 10 minutes to familiarize themselves with both the ultrasound equipment (SonoSite, MTurbo, Bothell, WA, USA) and the phantom model (MiniSim™ Upper Extremity Series, Life tech Inc., Stafford, Texas, USA). They also viewed a pre-recorded video demonstrating the task they were to perform. As a pre-test, participants performed the required Needle Insertion Accuracy (NIA) task 3 consecutive times and were assessed using a scoring form adapted from the Mayo Clinic. After completing the pre-test, participants were randomly divided into two groups, experimental and control, by a computer-generated randomization list (SAS Institute, Cary, NC). Participants were blinded to their group assignment.

Previously, we have reported details of the new learning tool. Briefly, all spatial movements occur in three dimensions which can be labeled the x-axis, the y-axis and the z-axis. A video camera records movement in two axes. By placing a second video camera at 90 degrees to the first camera, the third axis can be recorded as well as one axis in common with the first camera. Video recordings are stored electronically on a hard-drive and can be reviewed individually or in combination, at normal speed, or slowed if necessary. Still images can also be obtained.

The experimental group was allowed to practice the same pre-test task using the same ultrasound machine and phantom model. On a single computer screen, they were able to visualize their hand and needle movements along with the position of the ultrasound probe. The control group was allowed to practice the same pre-test task using the same ultrasound machine and phantom model but without the added visual aid. Both groups were allowed to practice their pre-test tasks for a maximum of 30 minutes, and recorded their self-assessment as proficient or not proficient at that time. Both groups then performed the post-test, which was the same task used for the pre-test, and each trainee was evaluated using the same scoring tool. To avoid subjective variations and inter-rater variability, all evaluations were recorded by a single blinded investigator.

Statistical analysis Pre- and post-test mean scores (ranging from 5 to15) were analyzed using statistical methods to determine whether this new learning tool improved NIA skills required with USRA. Pre-test and post-test scores (ranging from 5 to 15) were obtained in triplicate and averaged to produce a representative assessment for each participant. The primary endpoint was change in NIA score from baseline, i.e., the score difference obtained by subtracting the mean pre-test score from the mean post-test score. A sample size of 15 subjects per group (experimental and control) provides 80% power to detect an effect size of 1, based on a two-sided t-test with a 5% error probability (calculated using G*Power version 3.1). Analysis of the primary endpoint utilized a two-sided, two-sample t-test at the 5% level of significance. Secondary analyses evaluated the intervention effect on novice trainees, and trainees with prior USRA experience. Score differences for individual NIA skills (movement, alignment, approach, target, location) were also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Health Care professional

Exclusion Criteria:

* None

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Needle image accuracy score difference | 30 minutes
  The experimental group was allowed to practice the same pre-test task using the same ultrasound machine and phantom model. On a single computer screen, they were able to visualise their hand and needle movements along with the position of the ultrasound probe. The control group was allowed to practice the same pre-test task using the same ultrasound machine and phantom model but without the added visual aid. Both groups were allowed to practice their pre-test tasks for a maximum of 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Sanjib Adhikary, MB BS MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Result] Sites BD, Chan VW, Neal JM, Weller R, Grau T, Koscielniak-Nielsen ZJ, Ivani G. The American Society of Regional Anesthesia and Pain Medicine and the European Society of Regional Anaesthesia and Pain Therapy joint committee recommendations for education and training in ultrasound-guided regional anesthesia. Reg Anesth Pain Med. 2010 Mar-Apr;35(2 Suppl):S74-80. doi: 10.1097/AAP.0b013e3181d34ff5. PMID 20216029
- [Result] Ramlogan R, Manickam B, Chan VW, Liang L, Adhikary SD, Liguori GA, Hargett MJ, Brull R. Challenges and training tools associated with the practice of ultrasound-guided regional anesthesia: a survey of the American society of regional anesthesia and pain medicine. Reg Anesth Pain Med. 2010 Mar-Apr;35(2):224-6. doi: 10.1097/AAP.0b013e3181c69c94. No abstract available. PMID 20216042
- [Result] Adhikary SD, Hadzic A, McQuillan PM. Simulator for teaching hand-eye coordination during ultrasound-guided regional anaesthesia. Br J Anaesth. 2013 Nov;111(5):844-5. doi: 10.1093/bja/aet364. No abstract available. PMID 24108733
- [Result] Smith HM, Kopp SL, Jacob AK, Torsher LC, Hebl JR. Designing and implementing a comprehensive learner-centered regional anesthesia curriculum. Reg Anesth Pain Med. 2009 Mar-Apr;34(2):88-94. doi: 10.1097/AAP.0b013e31819e734f. No abstract available. PMID 19282705